CLINICAL TRIAL: NCT06629025
Title: The Clinical Manifestation and Prognosis of Pediatric Esophageal Motility Disorders
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202302017RIND
Record Dates: First submitted 2024-10-03; First posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2023-03

CONDITIONS: Esophageal Motility Disorders
Keywords: Esophageal achalasia; High-resolution esophageal manometry; Esophageal motility disorders in children
MeSH Terms: conditions — Esophageal Motility Disorders; Esophageal Achalasia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- esophageal motility disorder: Pediatric patients (0-20 years old) with clinically diagnosed abnormal esophageal motility
  Interventions: Diagnostic Test: High-resolution impedance manometry

INTERVENTIONS:
Diagnostic Test: High-resolution impedance manometry — High-resolution impedance manometry (HRIM) can calculate the bolus motion parameters and the ratio of complete esophageal transit
  Other Names: Peroral endoscopic myotomy (POEM)

SUMMARY:
Background: Abnormal esophageal peristalsis mostly occurs in adults, but some patients have onset in childhood. Most of the symptoms of esophageal motility disorders in children are not as clear as those described by adult patients, and they are only manifested in repeated vomiting. Esophageal peristalsis abnormalities in children took longer from symptoms to diagnosis than in adults. Common esophageal motility disorders in children include Achalasia, ineffective esophageal motility disorder (IEM), absent contractility, nutcracker esophagus, jackhammer esophagus, diffuse Esophageal spasm (diffuse esophageal spasm), lower esophageal sphincter hypertension (hypertensive lower esophageal sphincter), etc. Treatment for abnormal esophageal motility includes medication, endoscopic therapy, and surgery. This includes peroral endoscopic myotomy (POEM). The above treatment effects are rarely reported in children. This project uses the method of retrospective analysis of medical records to study the clinical manifestations and treatment prognosis of abnormal esophageal motility in children

Research purpose: The purpose of this study is to evaluate various clinical manifestations and treatment prognosis of abnormal esophageal motility in children, including analysis of diagnosis age, symptom time, related imaging examinations, endoscopy and high-resolution esophageal pressure examination, treatment methods, etc.

Research design: We plan to collect pediatric patients (0-20 years old) diagnosed with abnormal esophageal peristalsis at National Taiwan University Hospital during 2010/1/1-2022/12/31. Retrospective analysis of medical records and relevant laboratory data of patients in hospitals, including gender, height and weight, age of onset, symptoms, clinical manifestations, endoscopy, gastrointestinal photography, 24-hour multi-lumen esophageal impedance and acid-base examination, high-resolution esophageal pressure examination, ultrasound examination, pathological slide report, treatment response, etc.

Expected results: Analyze the clinical symptoms and different treatment methods of abnormal esophageal motility in children, and understand the development and prognosis of abnormal esophageal motility in children.

Key words: Esophageal motility disorders in children; High-resolution esophageal manometry; Esophageal achalasia

DETAILED DESCRIPTION:
1. Project name:

   The clinical manifestation and prognosis of pediatric esophageal motility disorders
2. Research purposes:

   The purpose of this study is to evaluate various clinical manifestations and treatment prognosis of esophageal motility disorders in children, including analysis of diagnosis age, symptom time, relevant imaging examinations, endoscopy and high-resolution esophageal pressure examination, treatment methods, etc.
3. Research background esophageal motility disorders occurs in adults, but there are still some patients with onset in childhood. Most of the symptoms of esophageal motility disorders in children are not as clear as those described by adult patients, and they are only manifested in repeated vomiting. Esophageal peristalsis abnormalities in children took longer from symptoms to diagnosis than in adults. Common esophageal motility disorders in children include Achalasia, ineffective esophageal motility disorder (IEM), absent contractility, nutcracker esophagus, jackhammer esophagus, diffuse Esophageal spasm (diffuse esophageal spasm), lower esophageal sphincter hypertension (hypertensive lower esophageal sphincter), etc. Treatment for abnormal esophageal motility includes medication, endoscopic therapy, and surgery. This includes peroral endoscopic myotomy (POEM). The above treatment effects are rarely reported in children. This project uses the method of retrospective analysis of medical records to study the clinical manifestations and treatment prognosis of abnormal esophageal motility in children
4. Participate in human research/clinical trials:

1. Main inclusion criteria: Pediatric patients (0-20 years old) who have been clinically diagnosed with abnormal esophageal motility 2. Main exclusion criteria: Exclude the diagnosis of abnormal esophageal motility

5. Research Design Pediatric patients (0-20 years old) who were diagnosed with esophageal motility disorders at National Taiwan University Hospital between January 1, 2010 and December 31, 2022. The medical records and relevant laboratory data of the patients at National Taiwan University Hospital were retrospectively analyzed, including Gender, height and weight, age of onset, symptoms, clinical manifestations, endoscopic examination, gastrointestinal photography, 24-hour multi-lumen esophageal impedance and acid-base examination, high-resolution esophageal pressure examination, ultrasound examination, pathological slide report, treatment response wait. During the data collection process, relevant medical records are stored in the Gastroenterology Laboratory of the Pediatric Department of National Taiwan University Hospital, which is locked. The computers and servers that store the data are protected by passwords. The data will be stored and analyzed in the hospital. Personal information that can be identified will be protected by code or file encryption. The host personally confirms that all researchers (including the host) have completed the training on medical record privacy protection and information security, and signed the conclusion of the confidentiality statement. When all the data is collected and analyzed, the moderator will completely de-identify the data.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients (0-20 years old) who have been clinically diagnosed with esophageal motility disorders

Exclusion Criteria:

* Exclude the diagnosis of esophageal motility disorders

Ages: 0 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: We plan to collect pediatric patients (0-20 years old) diagnosed with esophageal motility disorders at National Taiwan University Hospital during 2010/1/1-2022/12/31.
Sampling Method: Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2023-03-15 (Actual); Primary Completion 2024-02-05 (Actual); Study Completion 2024-02-05 (Actual)

PRIMARY OUTCOMES:
Treatment success rate of esophageal motility disorders | up to 10 years
Number of Patients with Serious and Non-Serious Adverse Events | up to 4 weeks
Time to Disease Progression | up to 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Chienting Hsu, Principal Investigator — 17F, No. 8, Chung-Shan South Rd, Taipei 100, Taiwan
Locations (1):
- National Taiwan University Children's Hospital, Taipei, Taiwan